CLINICAL TRIAL: NCT01621568
Title: A Phase II Study of Sunitinib in Patients With Advanced Relapsed or Refractory Thymoma or Thymic Carcinoma With at Least One Prior Line of Platinum-Based Systemic Chemotherapy
Brief Title: Sunitinib for Advanced Thymus Cancer Following Earlier Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120118; 12-C-0118
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Thymoma; Thymus Neoplasms
Keywords: VEGF; Anti-Angiogenesis; Targeted Agent
MeSH Terms: conditions — Thymoma; Thymus Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Thymoma and thymic carcinoma) (Experimental): Group 1 (Thymoma and thymic carcinoma) treated with sunitinib 50 mg/day, 4 weeks on, 2-weeks off (6 week cycle).
  Interventions: Drug: Sunitinib
- Group 2 (Thymic carcinoma only) (Experimental): Group 2 (Thymic carcinoma only) treated with sunitinib 50 mg/day, 2 weeks on, 1 week off (3 week cycle).
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50mg/day for 4 weeks daily, by mouth with 2 weeks off (6 week cycle)
  Other Names: Sutent
  Arms: Group 1 (Thymoma and thymic carcinoma)
Drug: Sunitinib — 50mg/day for 2 weeks daily, by mouth with 1 week off (3 week cycle)
  Other Names: Sutent
  Arms: Group 2 (Thymic carcinoma only)

SUMMARY:
Background:

- Sunitinib is drug that is approved for treating various types of cancers, including kidney cancers. However, it has not been approved to treat cancers of the thymus. Sunitinib works by blocking proteins that are responsible for cell division and growth. Some of these proteins can be found on thymus cancer cells. Researchers want to see if sunitinib can be used to treat advanced thymus cancer. It will be given to people who have had at least one earlier chemotherapy treatment containing platinum.

Objectives:

- To see if sunitinib is a safe and effective treatment for advanced thymus cancer that has not responded to earlier treatments.

Eligibility:

* Individuals at least 18 years of age who have advanced thymus cancer that has not responded to earlier treatments.
* At least one previous cancer treatment must have been chemotherapy treatment containing platinum.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and tumor biopsies will be used to check the severity of the cancer.
* Participants will take sunitinib tablets once a day, in the morning. They will take the tablets daily for 4 weeks, followed by 2 weeks of rest with no sunitinib. This 6-week period is called a cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Treatment cycles may be repeated as long as the tumor does not continue to grow and there are no severe side effects....

DETAILED DESCRIPTION:
BACKGROUND:

Platinum-based chemotherapy is the standard of care for advanced unresectable thymoma and thymic carcinoma. However over 50% of these patients may fail initial therapy and therefore require second-line therapy. New therapeutic options are needed for patients who have disease progression on or after platinum-containing therapy. Results obtained from protocol 12-C-0118 so far have shown impressive clinical activity of sunitinib in patients with recurrent thymic carcinoma with an objective response rate of 23% and disease control rate of 91% which is unprecedented for this histology. Treatment at a dose of 50 mg once daily for four weeks followed by 2 weeks off was poorly tolerated. Twenty five out of 41 patients needed dose reductions due to development of intolerable adverse events.

OBJECTIVES:

Primary objective:

- To evaluate the objective response rate (Partial Response (PR)+Complete Response (CR) for sunitinib in patients with relapsed or refractory thymoma or thymic carcinoma

MAIN ELIGIBILITY:

* Patients with histologically confirmed thymoma (Group 1 only) or thymic carcinoma who have previously been treated with at least one platinum-containing chemotherapy regimen with progressive disease prior to study entry
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Adequate renal, hepatic and hematopoietic function
* No major surgery, radiotherapy, chemotherapy or biologic therapy within 28 days of sunitinib

DESIGN:

* In the first group (Group 1), sunitinib will be administered orally using a continuous schedule at 50 mg per day for 4 weeks with 2 weeks off to constitute a 6-week cycle (Schedule 4/2) until disease progression or development of intolerable side-effects.
* In the second group (Group 2), sunitinib will be administered orally using a continuous schedule at 50 mg per day for 2 weeks with 1 week off to constitute a 3-week cycle (Schedule 2/1) until disease progression or development of intolerable side-effects.
* Toxicity will be assessed every cycle by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
* Tumor response assessments by RECIST 1.1 criteria will be performed every cycle for Group 1 and every other cycle for Group 2 (every 6 weeks) for patients receiving treatment for less than one year, and every two cycles for Group 1 and every four cycles for Group 2 (every 12 weeks) for patients who have been receiving treatment one year or longer.
* Exploratory studies include evaluation of serum vascular endothelial growth factor (VEGF), placental growth factor (PlGF), interleukin 4 (IL-4), interleukin 12 (IL-12), hepatocyte growth factor (HGF), and basic fibroblast growth factor (bFGF) (Group 1 only); and circulating tumor cells, endothelial progenitors, and mature apoptotic endothelial cells (both groups). In Group 2, regulatory T cells (Tregs), exhausted cluster of differentiation 8 (CD8) T cells, myeloid-derived suppressor cells (MDSCs), and Type 1 T helper (Th1)/Type 2 T helper (Th1) T cell populations will also be evaluated. Where tumor samples are available, intra-tumoral immune infiltrate will be assessed (both groups). Exploratory studies apply to National Cancer Institute (NCI) only.

ELIGIBILITY:
* INCLUSION CRITERIA:

3.1.1 Histological confirmation of thymoma (Group 1 only) or thymic carcinoma by the pathology department/Center for Cancer Research (CCR)/national Cancer Institute (NCI) or the pathology department of participating institutions.

3.1.2 At least one prior line of platinum-based chemotherapy or patient must have refused cytotoxic chemotherapy. Progressive disease must be documented prior to study entry.

3.1.3 Patients must not have received chemotherapy, radiation therapy, or undergone major surgery within 4 weeks prior to enrollment.

3.1.4 Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

3.1.5 Age greater than or equal to 18 years.

3.1.6 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky > 50 percent)

3.1.7 Life expectancy of greater than 3 months.

3.1.8 Patients must have normal organ and marrow function as defined below:

* hemoglobin greater than or equal to 9 g/dL
* leukocytes greater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,200/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin within normal institutional limits
* serum calcium less than or equal to 12.0 mg/dL
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT)/alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal
* creatinine within normal institutional limits

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
* If subjects have liver metastases, both ALT and AST must be less than or equal to 5 times upper limit of normal (ULN).
* Patients must have corrected QT Interval (QTc) < 500 msec

3.1.9 Prothrombin time (PT) or international normalized ratio (INR), and partial thromboplastin time test (APTT) less than or equal to 1.5 times upper limit of normal (ULN), unless the abnormality can be explained by the presence of lupus anticoagulant or if these values are in the therapeutic range for a patient on low molecular weight heparin.

3.1.10 The following groups of patients are eligible provided they have New York Heart Association Class II (NYHA) cardiac function on baseline echocardiogram (ECHO)/multi-gated acquisition scan (MUGA):

* those with a history of Class II heart failure who are asymptomatic on treatment
* those with prior anthracycline exposure
* those who have received central thoracic radiation that included the heart in the radiotherapy port.

3.1.11 Patients must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to study entry provided that the average of three BP readings at a visit prior to enrollment is less than 140/90 mmHg.

3.1.12 Absence of brain metastases as confirmed by imaging of the brain by magnetic resonance imaging (MRI) or computed tomography (CT) brain with contrast performed at baseline screening

3.1.13 The effects of sunitinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because anti-angiogenic agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of sunitinib administration.

3.1.14 Ability to understand and willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

3.2.1 Patients with tumor amenable to potentially curative therapy.

3.2.2 Prior treatment within the past 6 months with sunitinib, sorafenib, bevacizumab or other multikinase inhibitors targeting any of the following: vascular endothelial growth factors 1 3 (VEGF1 3), FMS-like tyrosine kinase 3 (FLT3), stem cell growth factor (c-KIT), platelet-derived growth factors-alpha and -beta (PDGF-alpha,-beta), colony-stimulating factor 1 (CSF1), and the RET receptor for glial-derived neurotrophic factors.

3.2.3 Patients with symptomatic brain metastases will be excluded from trial secondary to poor prognosis. However, patients who have had treatment for their brain metastasis and whose brain disease has remained stable for 3 months without steroid therapy may be enrolled.

3.2.4 Patients with evidence of severe or uncontrolled systemic disease, or any concurrent condition, which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies, uncontrolled hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection unless sustained virologic response to HCV therapy, uncontrolled diabetes, serious non-healing ulcer, wound or bone fracture, history of intra-abdominal abscess, abdominal fistula or gastrointestinal perforation within 28 days of treatment, history of pulmonary embolism in the past 12 months, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry, Class III or IV heart failure as defined by the NYHA functional classification system, stroke/cerebrovascular accident or transient ischemic attack within the past 12 months or psychiatric illness/social situations which would jeopardize compliance with the protocol.

3.2.5 History of a previous invasive malignancy within the last 5 years, except adequately treated non-melanoma skin cancer, papillary carcinoma of the thyroid or carcinoma in situ of the uterine cervix.

3.2.6 Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

3.2.7 Patients who are receiving any other investigational agents.

3.2.8 History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib. Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) are ineligible. (A list of potent CYP3A4 inducers or inhibitors can be found in Section 5.2.) An exception will be made for patients who are on ritonavir-based highly active antiretroviral therapy, in which case the starting dose of sunitinib will be modified as indicated in Sections 5.1.1 and 5.2.12. Every effort should be made to switch patients taking such agents or substances to other medications. A comprehensive list of medications and substances known or with the potential to alter the pharmacokinetics of sunitinib through CYP3A4 is provided.

3.2.9 Pregnant women are excluded from this study because sunitinib angiogenesis inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib breastfeeding should be discontinued if the mother is treated with sunitinib.

3.2.10 Patients who require therapeutic doses of Coumadin derivative anticoagulants such as warfarin are excluded. Low molecular weight heparin is permitted, provided the patient's prothrombin time (PT)/INR is less than or equal to 1.5. Coumadin doses of up to 2 mg daily are permitted for prophylaxis of thrombosis.

3.2.11 Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible.

3.2.12 Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded.

3.2.13 Patients with QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities are excluded.

3.2.14 Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 91 mmHg or higher) are ineligible.

3.2.15 Patients who require use of therapeutic doses of coumarin derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's PT INR is less than or equal to 1.5.

3.2.16 Patients with human immunodeficiency virus (HIV) infection are eligible provided their cluster of differentiation 4 (CD4) count is greater than or equal to the institutional lower limit of normal (LLN) ( greater than or equal to 334 cells/uL).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with study investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Detterbeck FC. Clinical value of the WHO classification system of thymoma. Ann Thorac Surg. 2006 Jun;81(6):2328-34. doi: 10.1016/j.athoracsur.2005.11.067. PMID 16731193
- [Background] Engels EA, Pfeiffer RM. Malignant thymoma in the United States: demographic patterns in incidence and associations with subsequent malignancies. Int J Cancer. 2003 Jul 1;105(4):546-51. doi: 10.1002/ijc.11099. PMID 12712448
- [Background] Falkson CB, Bezjak A, Darling G, Gregg R, Malthaner R, Maziak DE, Yu E, Smith CA, McNair S, Ung YC, Evans WK; Lung Cancer Disease Site Group of Cancer Care Ontario's Program in Evidence-Based Care. The management of thymoma: a systematic review and practice guideline. J Thorac Oncol. 2009 Jul;4(7):911-9. doi: 10.1097/jto.0b013e3181a4b8e0. PMID 19557895
- [Derived] Thomas A, Rajan A, Berman A, Tomita Y, Brzezniak C, Lee MJ, Lee S, Ling A, Spittler AJ, Carter CA, Guha U, Wang Y, Szabo E, Meltzer P, Steinberg SM, Trepel JB, Loehrer PJ, Giaccone G. Sunitinib in patients with chemotherapy-refractory thymoma and thymic carcinoma: an open-label phase 2 trial. Lancet Oncol. 2015 Feb;16(2):177-86. doi: 10.1016/S1470-2045(14)71181-7. Epub 2015 Jan 13. PMID 25592632
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0118.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2: Group 1 (Thymoma and thymic carcinoma) treated with sunitinib 50 mg/day, 4 weeks on, 2-weeks off (6 week cycle)
- No Treatment: Weeks 5-6, Group 1; Week 3, Group 2: Group 2 (Thymic carcinoma only) treated with sunitinib 50 mg/day, 2 weeks on, 1 week off (3 week cycle).
Period: Treatment Week 1-4
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2
Started | 41 | 15
Completed | 41 | 15
Not Completed | 0 | 0
Period: Week 5-6 No Treatment
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2
Started | 41 | 15
Completed | 39 | 15
Not Completed | 2 | 0
Not completed — Participant deemed ineligible and was taken off study. Did not receive treatment. | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2 | Total
Number analyzed (Participants) | 41 | 15 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 13 | 42
  >=65 years | 12 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.31 (11.35) | 58.67 (8.76) | 57.68 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 23 | 5 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 40 | 15 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 36 | 11 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 41 | 15 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response (Partial Response (PR) + Complete Response (CR) for Sunitinib in Participants With Relapsed or Refractory Thymoma or Thymic Carcinoma
Description: Objective response rate (CR + PR) will be measured according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria for sunitinib monotherapy in participants with advanced thymic malignancies. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: A median duration of 6 months
Population: 2/41 participants were not evaluable in group 1 thymoma and thymic carcinoma. 1/16 participants in group 2 thymic carcinoma were deemed ineligible and was taken off study. Did not receive treatment and was not assessed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1 (Thymoma Carcinoma) 50 mg/Day: Group 1 (Thymoma carcinoma) treated with sunitinib 50 mg/day, 4 weeks on, 2-weeks off (6 week cycle).
- Group 1 (Thymic Carcinoma) 50 mg/Day: Group 1 (Thymic carcinoma) treated with sunitinib 50 mg/day, 4 weeks on, 2-weeks off (6 week cycle).
- Group 2 (Thymic Carcinoma Only) 50 mg/Day: Group 2 (Thymic carcinoma only) treated with sunitinib 50 mg/day, 2 weeks on, 1 week off (3 week cycle).
Arm/Group | Group 1 (Thymoma Carcinoma) 50 mg/Day | Group 1 (Thymic Carcinoma) 50 mg/Day | Group 2 (Thymic Carcinoma Only) 50 mg/Day
Number analyzed (Participants) | 16 | 23 | 15
percentage of participants
  Complete Response | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Partial Response | 6 [0.2 to 30.2] | 26 [10.2 to 48.4] | 8 [0.2 to 36.0]

2. Secondary Outcome: Progression-free Survival for Sunitinib in Participants With Relapsed or Refractory Thymoma or Thymic Carcinoma
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesion, taking as reference the smallest sum on study; and the appearance of one or more new lesions.
Time Frame: An average of 10 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1 (Thymoma Carcinoma) 50 mg/Day | Group 1 (Thymic Carcinoma) 50 mg/Day | Group 2 (Thymic Carcinoma Only) 50 mg/Day
Number analyzed (Participants) | 16 | 23 | 15
Months | 8.5 [2.8 to 11.3] | 7.2 [3.4 to 15.2] | 5.0 [2.7 to 5.5]

3. Secondary Outcome: Number of Participants Alive at 1 Year After Treatment With Sunitinib
Description: Number of participants alive at 1 year after treatment with sunitinib.
Time Frame: 12 months after initiation of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Thymoma Carcinoma) 50 mg/Day | Group 1 (Thymic Carcinoma) 50 mg/Day | Group 2 (Thymic Carcinoma Only) 50 mg/Day
Number analyzed (Participants) | 16 | 23 | 15
Participants | 14 | 18 | 9

4. Secondary Outcome: Number of Grades ≥3 Adverse Events Related to Sunitinib
Description: Adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 110 months and 28 days for the thymoma/thymic carcinoma group and 91 months and 11 days for the thymic carcinoma only group.
Population: For toxicity, histology does not make a difference and tolerability is dependent on the schedule. Hence, we combined the two parts of group 1 (thymoma and thymic carcinoma) and reported the data in two groups.
Measure: Number; unit: Adverse events
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2
Number analyzed (Participants) | 41 | 15
Adverse events
  Grade 3 | 95 | 40
  Grade 4 | 6 | 3
  Grade 5 | 1 | 0

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 4
Population: 1/16 participants in the thymic group were deemed ineligible and was taken off study. Did not receive treatment and was not assessed for adverse events. For toxicity, histology does not make a difference and tolerability is dependent on the schedule. Hence, we combined the two parts of group 1 (thymoma and thymic carcinoma) and reported the data in two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2
Number analyzed (Participants) | 41 | 15
Participants | 41 | 15

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 110 months and 28 days for the thymoma/thymic carcinoma group and 91 months and 11 days for the thymic carcinoma only group.
Description: 1/16 participants in the thymic group were deemed ineligible and was taken off study. Did not receive treatment and was not assessed for adverse events. For toxicity, histology does not make a difference and tolerability is dependent on the schedule. Hence, we combined the two parts of group 1 (thymoma and thymic carcinoma) and reported the data in two groups.
Arm/Group | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2
All-Cause Mortality (participants affected / at risk) | 38/41 | 15/15
Serious Adverse Events (participants affected / at risk) | 38/41 | 15/15
Other Adverse Events (participants affected / at risk) | 40/41 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 (N=41) | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2 (N=15)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Death NOS (General disorders) | 38 (38) | 15 (15)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) — Death due to progressive disease
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Weeks 1-4, Group 1; Weeks 1-2, Group 2 (N=41) | No Treatment: Weeks 5-6, Group 1; Week 3, Group 2 (N=15)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 2 (5)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 20 (35) | 2 (4)
Alkaline phosphatase increased (Investigations) | 13 (17) | 2 (3)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 28 (87) | 4 (9)
Anorexia (Metabolism and nutrition disorders) | 21 (27) | 7 (11)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 27 (58) | 4 (5)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 11 (18) | 1 (2)
Blurred vision (Eye disorders) | 4 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CPK increased (Investigations) | 2 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 7 (7) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (16) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 5 (8)
Creatinine increased (Investigations) | 4 (5) | 3 (31)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (4)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 24 (60) | 10 (18)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 17 (26) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 17 (22) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 3 (6)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 8 (13) | 2 (2)
Edema limbs (General disorders) | 11 (13) | 3 (4)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 4 (6) | 2 (2)
Endocrine disorders - Other, Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, Low testosterone (Endocrine disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Eye disorders - Other, Ptosis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Floaters (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Light sensitivity (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Puffy eyes (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Right eye subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Right eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Visual changes (Eye disorders) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 31 (79) | 7 (9)
Fever (General disorders) | 8 (8) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (12) | 2 (2)
Gastrointestinal disorders - Other, Black stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Mouth Sore (Gastrointestinal disorders) | 1 (4) | 0 (0)
Gastrointestinal disorders - Other, Sore mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Whole body edema (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (14) | 1 (2)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 4 (5) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (11) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (17) | 1 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Hypertension (Vascular disorders) | 17 (21) | 4 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 (56) | 6 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (10) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (12) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 10 (12) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (21) | 4 (6)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 9 (10) | 2 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Infections and infestations - Other, Finger (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Flu (Infections and infestations) | 2 (2) | 0 (0)
Infections and infestations - Other, Nose Wound (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Oral Infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Sinus (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Infections and infestations - Other, Thrush (Infections and infestations) | 2 (3) | 0 (0)
Infections and infestations - Other, face, eye (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 25 (114) | 9 (60)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 23 (44) | 8 (17)
Musculoskeletal and connective tissue disorder - Other, Finger Cracking (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Hand Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Plantar Fasciitis Left foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nail loss (Infections and infestations) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 22 (32) | 8 (12)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Gastric polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Other, Bilateral feet (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Other, Heat sensitivity (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Mild numbness left lower jaw and chin (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Wrist Drop (Nervous system disorders) | 1 (3) | 0 (0)
Nervous system disorders - Other, dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 25 (65) | 6 (25)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 10 (14) | 4 (5)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 7 (17) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (9) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 (30) | 5 (10)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Periorbital edema (Cardiac disorders) | 1 (1) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (10) | 2 (2)
Platelet count decreased (Investigations) | 25 (66) | 10 (34)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary valve disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (10) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Bloody Stools (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, Rectal Bleeding (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 9 (9) | 1 (1)
Sinusitis (Infections and infestations) | 5 (10) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Changes color (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Color change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Facial Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hair hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Itching (anus) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Perianal rash. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash (rectal/anus) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash- feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, change of hair color (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Yellowing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Yellowing of palms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, nail cracking (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Yellow skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 6 (7) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (26) | 4 (8)
Watering eyes (Eye disorders) | 1 (1) | 1 (1)
Weight gain (Investigations) | 2 (6) | 0 (0)
Weight loss (Investigations) | 5 (7) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 26 (100) | 10 (72)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT01621568/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Standard Group 1 Consent (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT01621568/ICF_001.pdf
  • Informed Consent Form: Standard Group 2 Consent (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT01621568/ICF_003.pdf